CLINICAL TRIAL: NCT02176408
Title: Efficacy of Adjunctive Exercise for the Behavioral Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F31MH100773-01A1 (NIH); F31MH100773-01A1 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; MDD; Exercise; Physical Activity; Treatment; Behavioral Activation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Activation plus Exercise (Experimental): Six weekly 60-minute sessions plus three 60-minute biweekly booster sessions of behavioral activation treatment
  Six weekly 30-minute sessions of the exercise intervention (with this intervention incorporated into the 60 minutes of the biweekly booster sessions)
  Interventions: Behavioral: Behavioral Activation; Behavioral: Exercise Intervention
- Behavioral Activation plus Stretching (Active Comparator): Six weekly 60-minute sessions plus three 60-minute biweekly booster sessions of behavioral activation treatment
  Six weekly 30-minute sessions of the stretching intervention (with this intervention incorporated into the 60 minutes of the biweekly booster sessions)
  Interventions: Behavioral: Behavioral Activation; Behavioral: Stretching Intervention

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral Activation Therapy (BA). All participants will receive a standard behavioral activation treatment based on the manualized treatment described by Lejuez et al., 2011. Treatment will be delivered in 60-minute weekly sessions over a 6-week period followed by 3 biweekly booster sessions. Behavioral activation includes scheduling activities the patient will enjoy and find important with the purpose of improving mood.
Behavioral: Exercise Intervention — Exercise Intervention (EX). The exercise intervention will immediately follow each of the first six weekly BA sessions. Each EX session will comprise 30 minutes of either providing rationale for the program or reviewing the previous week's progress. As part of the intervention, participants will be asked to perform 40 minutes of aerobic exercise at 60-75% of maximum heart rate on three days each week, with 5 minute stretching warm up and cool down. We will help all participants initiate and plan their at-home program of exercise.
  Arms: Behavioral Activation plus Exercise
Behavioral: Stretching Intervention — Stretching Intervention (STR). The stretching intervention will also follow each of the first six weekly BA sessions. These sessions will comprise 30 minutes of providing rationale for the stretching program or reviewing the previous week's progress. As part of the intervention, participants will be asked to perform 50 minutes of stretching on three days each week. Participants in this condition will be provided with a 50-minute DVD of stretching exercises and will work with the therapist to plan their at-home stretching exercises.
  Arms: Behavioral Activation plus Stretching

SUMMARY:
Major depressive disorder (MDD) is the leading cause of disability in the developed world and is associated with lost productivity, increased health care utilization, and mortality. Several empirically supported treatments, such as antidepressant medication and cognitive behavioral therapy, exist for the treatment of MDD; however, studies have shown that as many as 34% of individuals do not respond to these treatments. Exercise and stretching interventions represent alternative strategies associated with strong effect sizes in past studies. Additionally, exercise has been shown to enhance cognitive functioning, especially attention and memory. This study aims to investigate the effect of a combined aerobic exercise and behavioral activation treatment (BA) for MDD. Behavioral activation treatment involves completing both pleasant and mastery-based activities with the goal of enhancing mood. The current study will recruit 32 MDD patients for an active treatment phase of nine 60-90 minute sessions (6 weekly sessions and 3 biweekly sessions) of either BA plus exercise (BA+EX) or BA plus stretching (BA+STR). The purpose of this study is to identify if adding aerobic exercise to a brief psychosocial treatment can improve mood above and beyond an active control condition.

DETAILED DESCRIPTION:
Individuals with major depressive disorder (MDD) will be recruited to participate in a free treatment trial of a combined exercise or stretching regimen plus behavioral activation treatment. All individuals will receive 6 weekly and 3 biweekly 1-hour sessions of behavioral activation treatment. Behavioral activation involves exploring values in different life areas (relationships, education/career, interests, etc.) and scheduling activities in line with these values. Research has shown that behavioral activation treatment can improve mood and alleviate depressive symptoms.

In addition, participants will be randomized (like a flip of a coin) to either an additional aerobic exercise intervention or an additional stretching intervention. These interventions will take place for half an hour after the first 6 weeks of the behavioral activation intervention. The purpose of this study is to examine if adding an aerobic exercise intervention to a brief psychosocial treatment can improve mood above and beyond an active control condition.

Throughout the study, participants will complete computer, questionnaire, and interview assessments as well as exercise tests and a blood draw. The details of each visit are listed below. For full completion of this study, participants can earn up to $100.

Screening visit: diagnostic interview, assessment for physical activity risk (brief meeting with physician)

Baseline visit (week 0): submaximal exercise test, blood draw, questionnaire measures, computer tests

Treatment visit 1 (week 1): BA treatment + EX/STR intervention, brief questionnaires

Treatment visit 2 (week 2): BA treatment + EX/STR intervention, brief questionnaires

Treatment visit 3 (week 3): BA treatment + EX/STR intervention, brief questionnaires

Treatment visit 4 (week 4): BA treatment + EX/STR intervention, questionnaires, submaximal exercise test, blood draw

Treatment visit 5 (week 5): BA treatment + EX/STR intervention, brief questionnaires

Treatment visit 6 (week 6): BA treatment + EX/STR intervention, brief questionnaires

Treatment visit 7 (week 8): BA treatment, questionnaires, submaximal exercise test, blood draw

Treatment visit 8 (week 10): BA treatment, brief questionnaires

Treatment visit 9 (week 12): BA treatment, questionnaire measures

Final assessment (week 16): submaximal exercise test, blood draw, questionnaire measures, computer tests

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-65 with a principal DSM-5 diagnosis of MDD or Persistent Depressive Disorder with a current Major Depressive Episode (as determined by the Anxiety and Related Disorders Interview Schedule-5)
* Sedentary (moderate-intensity exercise less than two days per week for at least 30 minutes each time for at least 3 months)
* Able to provide informed consent for the study
* Sufficient command of the English language

Exclusion Criteria:

* Current or past psychotic disorders of any type, bipolar disorder (I, II, or NOS), schizophrenia or schizoaffective disorder, anorexia, bulimia, or alcohol or drug dependence
* Currently suicidal or high suicide risk (as evaluated by the Columbia Suicide Severity Rating Scale and BDI suicide item)
* Risk for exercise according to the Physical Activity Readiness Questionnaire (PAR-Q) in accordance with the guidelines set forth by the American College of Sports Medicine (ACSM) (i.e., existence of the conditions in the next bullet point)
* Physical conditions (e.g.,heart conditions, diabetes, asthma or another lung disease, bone/joint problems, or seizure disorder) interfering with the ability to exercise safely
* Individuals who have participated in cognitive behavioral therapy (CBT) directed towards the treatment of a mood disorder within three months of baseline, those simultaneously participating in another psychosocial treatment (other than supportive therapy) or those not currently stable (i.e., same dosage for at least 8 weeks) on psychotropic medications
* Women who are currently pregnant, plan to be pregnant in the next year, or currently breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Szuhany, M.A., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Szuhany KL, Otto MW. Assessing BDNF as a mediator of the effects of exercise on depression. J Psychiatr Res. 2020 Apr;123:114-118. doi: 10.1016/j.jpsychires.2020.02.003. Epub 2020 Feb 8. PMID 32065946
- [Derived] Szuhany KL, Otto MW. Efficacy evaluation of exercise as an augmentation strategy to brief behavioral activation treatment for depression: a randomized pilot trial. Cogn Behav Ther. 2020 May;49(3):228-241. doi: 10.1080/16506073.2019.1641145. Epub 2019 Jul 30. PMID 31357916

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven participants were enrolled in the study but not randomized to one of the two intervention arms. Four participants were excluded after the screening visit due to not meeting study inclusion criteria. Three participants completed screening but discontinued the study prior to attending the baseline visit (during which randomization occurs).
Groups:
- Behavioral Activation Plus Exercise: Six weekly 60-minute sessions plus three 60-minute biweekly booster sessions of behavioral activation treatment
  Six weekly 30-minute sessions of the exercise intervention (with this intervention incorporated into the 60 minutes of the biweekly booster sessions)
  Behavioral Activation Therapy (BA). All participants received standard BA based on the manualized treatment described by Lejuez et al., 2011. BA includes scheduling activities the patient will enjoy and find important with the purpose of improving mood.
  Exercise Intervention (EX). Each EX session had 30 minutes of either providing rationale for the program, reviewing motivational strategies, or reviewing the previous week's progress.
- Behavioral Activation Plus Stretching: Six weekly 60-minute sessions plus three 60-minute biweekly booster sessions of behavioral activation treatment
  Six weekly 30-minute sessions of the stretching intervention (with this intervention incorporated into the 60 minutes of the biweekly booster sessions)
  Behavioral Activation Therapy (BA). All participants received standard BA based on the manualized treatment described by Lejuez et al., 2011. BA includes scheduling activities the patient will enjoy and find important with the purpose of improving mood.
  Stretching Intervention (STR). These sessions had 30 minutes of providing rationale for the stretching program, reviewing motivational strategies, or reviewing the previous week's progress.
Period: Overall Study
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Started | 15 | 16
Completed | 9 | 12
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (12.7) | 36.5 (13.7) | 34.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item clinician-rated measure of correlates of depression. Specifically, this questionnaire measures the following: sadness, tension, sleep, appetite, concentration, lassitude, numbness, pessimism, and suicidal ideation. The scale ranges from 0-60 with higher totals indicating worse depression. The following are norms for severity: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; and >34 - severe depression.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 11.2 (7.5) | 16.0 (9.5)

2. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The BDI is a widely used 21-item, self-report inventory designed to measure severity of depressive symptoms. Scores range from 0-63 with higher scores indicating worse depression. The following are severity norms for the measure: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 8.7 (9.5) | 13.2 (9.6)

3. Secondary Outcome: Work and Social Adjustment Scale (WSAS)
Description: The WSAS is a self-report scale of functional impairment attributable to an identified problem, in this case MDD. Scores range from 0 to 40 with higher scores indicating worse functioning. A WSAS score above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinicalsymptomatology. Scores below 10 appear to be associated with subclinical populations.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 10.7 (10.5) | 16.5 (12.5)

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Q-LES-Q rates 16 aspects of quality of life, including physical health, mood, activities of daily living, and overall life satisfaction. Scores range from 14 to 70 with lower scores indicating worse quality of life.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 53.9 (9.0) | 45.5 (10.6)

5. Secondary Outcome: Logical Memory
Description: Participants will be read a story and asked to remember as many details as possible. Raw scores are reported with a range in the current sample from from 17 to 47 with higher scores indicating better memory performance.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 34.75 (10.54) | 28.18 (6.29)

6. Secondary Outcome: Continuous Performance Test- Identical Pairs
Description: Participants' attention will be assessed using the CPT which is a choice reaction time task which requires a subject to respond whenever two identical stimuli appear in a row within a sequence of rapidly flashed trials. Scores represent the average d' across 2 digit, 3 digit, and 4 digit trials. Average scores in this sample ranged from 1.76 to 4.24. Lower d' represents a better score.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
score on a scale | 2.99 (.41) | 3.05 (.66)

7. Secondary Outcome: 7 Day Physical Activity Recall (PAR)
Description: The PAR is is an interviewer-administered measure of physical activity behavior that will be used as a self-report validation measure of amount of physical activity completed. Metabolic equivalents (METs) of moderate and vigorous intensity activity are reported. METs of activity ranged from 0 to 1520 in this sample with higher numbers indicating more physical activity completed.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: METs
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 15 | 16
METs | 752.89 (447.57) | 530.00 (515.01)

8. Secondary Outcome: Brain-derived Neurotrophic Factor (BDNF)
Description: Blood samples (approximately 1 tsp) will be collected at baseline, week 4, week 8, and week 16 to test serum BDNF. Changes in resting BDNF levels were assessed. BDNF levels ranged from 14391 to 43020 ng/ml in this sample with higher levels indicating more BDNF.
Time Frame: Week 16
Population: Amount of individuals who had BDNF data available at Week 16.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
Number analyzed (Participants) | 7 | 9
ng/mL | 25996.86 (3807.37) | 26601.11 (9237.28)

ADVERSE EVENTS:
Time Frame: Collected over the course of the entire study (16 weeks per participant)
Arm/Group | Behavioral Activation Plus Exercise | Behavioral Activation Plus Stretching
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/16
Other Adverse Events (participants affected / at risk) | 1/15 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation Plus Exercise (N=15) | Behavioral Activation Plus Stretching (N=16)
Inpatient hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — 1 day inpatient hospitalization for suicidal ideation
Inpatient hospitalization (Social circumstances) | 0 (0) | 1 (1) — 4 day inpatient hospitalization for excessive alcohol consumption
Inpatient hospitalization (General disorders) | 1 (1) | 0 (0) — Inpatient hospitalization due to dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation Plus Exercise (N=15) | Behavioral Activation Plus Stretching (N=16)
Sprained ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (5)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study had limited power to detect overall treatment differences given higher levels of dropout than expected, had limited follow-up, and a lack of a waitlist (or no movement) control condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No